CLINICAL TRIAL: NCT05865626
Title: A Pilot Study to Evaluate Video Observed Treatment Among Tuberculosis Patients From Lambaréné Using an Instant Messenger Application
Brief Title: Evaluation of the VOT Among Tuberculosis Patients From Lambaréné
Acronym: dotsapp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Responsible Party: Principal Investigator, EDOA Jean Ronald, Dr, Centre de Recherche Médicale de Lambaréné
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: dotsapp1
Record Dates: First submitted 2023-04-29; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: In the intervention group, 20 subjects will receive a smartphone and one of the two incentives (close-follow-up or a financial incentive) over a 12 weeks period. After this period, the participant will receive the second incentive. The order is determined randomly with 10 participants receiving the incentives. Participants may receive a third incentive (social feedback) the earliest 6 weeks after the beginning of the treatment, in addition to the basic incentive. The 10 participants in the control group will not receive a smartphone but will be followed-up monthly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VOT without cash incentive at the begining (Experimental): Participants in this group start VOT without financial motivation. In the second part of their follow-up, VOT is combined with financial motivation.
  Interventions: Other: VOT with and without cash incentive
- VOT with cash incentive at the begining (Experimental): The participants in this group start the VOT with the financial motivation. In the second part of their follow-up, VOT is no longer associated with financial motivation
  Interventions: Other: VOT with and without cash incentive
- Standard care (No Intervention): The participants in this group self-administer the anti-tuberculosis treatment as is done routinely.

INTERVENTIONS:
Other: VOT with and without cash incentive — Here we are interested in the remote monitoring of TB treatment, and the impact that financial motivation can have on compliance with this monitoring. the cross-over here means that participants in each intervention group will at some point receive VOT without motivation and then VOT with motivation, depending on whether they start with one or the other combination
  Other Names: VOT
  Arms: VOT with cash incentive at the begining; VOT without cash incentive at the begining

SUMMARY:
This pilot study aimed to assess the feasibility of using an instant messenger to monitor drug intake in tuberculosis patients and to assess cash incentive to improve adherence to drug intake

DETAILED DESCRIPTION:
At the initial visit, the inclusion criteria are cross-checked, the subject is informed of the study procedures, and an informed consent form is signed by subjects willing to participate.

For the participants from the intervention group, the research team will provide a smartphone with the WhatsApp application to each participant. At the initial visit, the research team will explain to the participants how to use the phone and the instant messenger application for the study. Briefly, the subject is filmed while taking the drug. This can be via a "selfie" or by a family member. The video is then sent to the study phone contact.

Once the video is received by an investigator, a message will be sent back to the participant's mobile phone acknowledging receipt of the video. An investigator trained on the DOT protocol, will review the video clips to assess if the drug was taken correctly or not. A daily log is filled in to keep track of drug intake for each participant.

Participants from both the control and intervention group are seen once per month in person for follow-ups and getting new drugs. At these time points information on drug intake is gathered.

ELIGIBILITY:
Inclusion Criteria:

Older than 18 years

* Signed informed consent form
* Living in an area with mobile phone coverage
* Have at least 3 months of treatment remaining

Exclusion Criteria:

• Not being able to use a smartphone and unlikely to learn how to

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
feasibility assessment | at the end of study (2 years)
  proportion of participants in the intervention groups who regularly send the videos throughout the follow-up.

SECONDARY OUTCOMES:
adherence to the VOT | at the end of study (2 years)
  number of videos received compared to the expected number of videos
effect of cash incentives on adherence to the VOT | at the end of study (2 years)
  comparison of the proportion of videos received during the follow-up phase without financial motivation and the proportion of videos received during the follow-up phase with financial motivation.

CONTACTS AND LOCATIONS:
Overall Officials: Bertarnd Lell, prof., Study Director — Centre de Recherche Médicale de Lambaréné
Locations (1):
- Centre de recherches médicales de Lambaréné, Lambaréné, Gabon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belard S, Remppis J, Bootsma S, Janssen S, Kombila DU, Beyeme JO, Rossatanga EG, Kokou C, Osbak KK, Obiang Mba RM, Kaba HM, Traore AN, Ehrhardt J, Bache EB, Flamen A, Rusch-Gerdes S, Frank M, Adegnika AA, Lell B, Niemann S, Kremsner PG, Loembe MM, Alabi AS, Grobusch MP. Tuberculosis Treatment Outcome and Drug Resistance in Lambarene, Gabon: A Prospective Cohort Study. Am J Trop Med Hyg. 2016 Aug 3;95(2):472-80. doi: 10.4269/ajtmh.15-0668. Epub 2016 Jun 27. PMID 27352879
- [Background] Elangovan R, Arulchelvan S. A Study on the Role of Mobile Phone Communication in Tuberculosis DOTS Treatment. Indian J Community Med. 2013 Oct;38(4):229-33. doi: 10.4103/0970-0218.120158. PMID 24302824
- [Background] Sinkou H, Hurevich H, Rusovich V, Zhylevich L, Falzon D, de Colombani P, Dadu A, Dara M, Story A, Skrahina A. Video-observed treatment for tuberculosis patients in Belarus: findings from the first programmatic experience. Eur Respir J. 2017 Mar 22;49(3):1602049. doi: 10.1183/13993003.02049-2016. Print 2017 Mar. PMID 28331042
- [Background] Garfein RS, Collins K, Munoz F, Moser K, Cerecer-Callu P, Raab F, Rios P, Flick A, Zuniga ML, Cuevas-Mota J, Liang K, Rangel G, Burgos JL, Rodwell TC, Patrick K. Feasibility of tuberculosis treatment monitoring by video directly observed therapy: a binational pilot study. Int J Tuberc Lung Dis. 2015 Sep;19(9):1057-64. doi: 10.5588/ijtld.14.0923. PMID 26260824
- [Background] Handbook for the use of digital technologies to support tuberculosis medication adherence. Geneva: World Health Organization; 2017.
- [Background] Iribarren SJ, Schnall R, Stone PW, Carballo-Dieguez A. Smartphone Applications to Support Tuberculosis Prevention and Treatment: Review and Evaluation. JMIR Mhealth Uhealth. 2016 May 13;4(2):e25. doi: 10.2196/mhealth.5022. PMID 27177591
- [Background] Giordano V, Koch H, Godoy-Santos A, Dias Belangero W, Esteves Santos Pires R, Labronici P. WhatsApp Messenger as an Adjunctive Tool for Telemedicine: An Overview. Interact J Med Res. 2017 Jul 21;6(2):e11. doi: 10.2196/ijmr.6214. PMID 28733273
- [Background] Seewoodharry MD, Maconachie GDE, Gillies CL, Gottlob I, McLean RJ. The Effects of Feedback on Adherence to Treatment: A Systematic Review and Meta-analysis of RCTs. Am J Prev Med. 2017 Aug;53(2):232-240. doi: 10.1016/j.amepre.2017.03.005. Epub 2017 Apr 26. PMID 28456347
- [Background] Lutge EE, Wiysonge CS, Knight SE, Sinclair D, Volmink J. Incentives and enablers to improve adherence in tuberculosis. Cochrane Database Syst Rev. 2015 Sep 3;2015(9):CD007952. doi: 10.1002/14651858.CD007952.pub3. PMID 26333525
- [Background] Stuurman AL, Vonk Noordegraaf-Schouten M, van Kessel F, Oordt-Speets AM, Sandgren A, van der Werf MJ. Interventions for improving adherence to treatment for latent tuberculosis infection: a systematic review. BMC Infect Dis. 2016 Jun 8;16:257. doi: 10.1186/s12879-016-1549-4. PMID 27268103